CLINICAL TRIAL: NCT04141488
Title: Examining The Efficacy Of Scapular Exercises On Pain, Muscle Activation And Function İn Patients With Lateral Epicondylitis
Brief Title: Examining The Efficacy Of Scapular Exercises On Pain And Function İn Patients With Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Bayram Kapşigay, Research Assistant, Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BitlisErenU
Record Dates: First submitted 2019-10-16; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Lateral Epicondylitis
Keywords: Lateral Epicondylitis; electromyography; pain; scapula
MeSH Terms: conditions — Tennis Elbow; Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimantel Group (Experimental): Electrotherapy program in our study 20 minutes, Hot-pack (HP) 20 minutes, 60-120 Hz frequency range 50-100 millisecond pulse time conventional TENS (Transcutaneous Electrical Nerve Stimulation) and 5 minutes 1.5 watt / cm2 treatment dosage 1 MHz ' ultrasound (US) treatment was applied. Exercise program; Eccentric and concentric strengthening and stretching of ECBR and ECBL muscles, terminal elbow flexion and extension, forearm pronation and supination exercises were given. Electrotherapy was given as 15 sessions for 6 weeks, 2 or 3 days a week, 1 session per day, and 30 sessions for 6 weeks, 5 days per week. Fifteen of these exercise sessions were supervised by the physiotherapist in the hospital and the remaining 15 patients did not come to the clinic on their own. The experimantel group was given strengthening exercises of the upper trapezoidal, middle trapezoidal and serratus anterior muscles with extra scapula muscles.
  Interventions: Other: experimantal group
- Control Group (Other): Electrotherapy program in our study 20 minutes, Hot-pack (HP) 20 minutes, 60-120 Hz frequency range 50-100 millisecond pulse time conventional TENS (Transcutaneous Electrical Nerve Stimulation) and 5 minutes 1.5 watt / cm2 treatment dosage 1 MHz ' ultrasound (US) treatment was applied. Exercise program; Eccentric and concentric strengthening and stretching of ECBR and ECBL muscles, terminal elbow flexion and extension, forearm pronation and supination exercises were given. Electrotherapy was given as 15 sessions for 6 weeks, 2 or 3 days a week, 1 session per day, and 30 sessions for 6 weeks, 5 days per week. Fifteen of these exercise sessions were supervised by the physiotherapist in the hospital and the remaining 15 patients did not come to the clinic on their own.
  Interventions: Other: experimantal group

INTERVENTIONS:
Other: experimantal group — Control Group
  Other Names: Control Group

SUMMARY:
We aimed to investigate the effect of scapular exercises on pain and functioning in patients with lateral epicondylitis to achieve a more accurate result by using little-used EMG between scapula and elbow muscles in the literature besides ongoing classical measurements and evaluations.

DETAILED DESCRIPTION:
Thirty patients who participated in the study were randomly divided into two groups. First group (n=15), conventional physiotherapy program and exercise, second group (n=15), in addition to the conventional physiotherapy program and exercises, scapula exercises were applied. Patients were evaluated before and after treatment by VAS, algometer, hand dynamometer, EMG, UEFS, PRTEE and DASH questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Cases diagnosed with lateral epicondylitis by the physician and decided to receive conservative treatment
* Not receiving NSAID or other medical treatment
* Untreated Lateral Epicondylitis for the last 6 months
* Cases with age range 18-75
* Patients with pain and tenderness for at least 3 months

Exclusion Criteria:

* People with pacemakers or cardiac arrhythmias
* Tumoral disease
* Pregnant women
* Head and neck, elbow, scapula joint pathologies
* Acute infection
* Nerve or nerve root compression
* Other musculoskeletal problems

Ages: 25 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Pain Severity Assessment | Change from baseline pain severity of Lateral Epicondylitis at week 6.
  In order to evaluate the general pain severity of the patients, Visual Analog Scale (VAS), which is the Visual Pain Scale of Turkish, was used. Patients were asked to mark their general pain separately on a 10 cm scale. According to this, "0" indicates that there is no pain, and "10" indicates the most severe pain. The distance between the marked point and the beginning of the line was recorded in centimeters
Muscle Activation Assessment | Change from baseline EMG activation of the forearm extensor muscles at week 6.
  In order to record the EMG signals of the ECRB muscle, the bipolar Ag / AgCl was adhered to the designated area at a distance of 1 cm between the centers of the superficial electrodes according to SENİAM criteria and the reference electrode was placed in the farthest region. Before the electrodes were bonded, the skin surface was shaved with a razor blade and cleaned with isopropyl alcohol to get a better signal. The measurements were made simultaneously in grip position with the automatically tuned EMG biofeedback.
Functional Level Assessment | Change from baseline functional level score at week 6.
  In order to determine the level of functional, "Arm, Shoulder and Hand Problems Questionnaire (DASH-T)" was used. The scale consists of three parts. The first 21 questions assess the patient's difficulty during daily life activities, 5 questions assess symptoms (pain, pain due to activity, tingling, stiffness, weakness), and the remaining 4 questions assess social function, work, sleep and self-confidence. Each question is scored from 1 to 5 and subtracted from 1, multiplied by 25. A high score indicates a bad apology.
Functionality Assessment | Change from baseline functionality score at week 6.
  In order to measure yhe functionality Upper Extremity Functionality Indeks (UEFI) was used. It consists of 8 questions. These include questions such as opening jars, driving more than 30 minutes, sleeping, writing, grasping small objects with their fingers, taking jugs from the refrigerator, opening doors and washing dishes. A visual scale is asked for each question. 1 shows that there is no pain and 10 indicates that the pain is the most severe. The total score is between 8-80.

SECONDARY OUTCOMES:
Grip Force Assessment | Change from baseline grip force score at week 6.
  Grip force was made by JAMAR brand dynamometer. The first measurement was performed with the elbow 90o flexed in the sitting position, the forearm in the neutral position, the shoulder adduction, the wrist between 0-30o and arm supported in the chair, the second measurement was repeated averaged five times while the arm was in adduction in the elbow extension, and the mean was recorded in terms of (lbs) -force.
Pressure Pain Threshold Assessment | Change from baseline Pressure Pain Threshold score at week 6.
  It is a device used to evaluate pain sensitivity and to determine pressure perception. The pressure pain threshold is defined as the minimum pressure that causes pain or discomfort. In our study, pressure gauge res J Tech Commander Algometer produced by "J Tech Medical" was used to determine the pressure pain threshold. The device is a digital pain threshold meter and consists of a sensor connected to the hard tip with a diameter of 1 cm. The measurement was performed in sitting position, shoulder abduction, elbow, forearm, wrist and hand. Patients were previously told to stop the therapist at the point where the pressure turned into a painful sensation and continued to the limit that the patient could withstand by applying a compressive pressure on the lateral epicondyle

CONTACTS AND LOCATIONS:
Overall Officials: Bayram Kapsigay, MSc, Principal Investigator — Bitlis Eren University
Locations (2):
- Turkey (Türkiye) (2):
  - Bayram Kapsigay, Istanbul, Maltepe
  - Marmara University, Istanbul